CLINICAL TRIAL: NCT03237845
Title: BHV3000-302 : Phase 3: Double-Blind, Randomized, Placebo-Controlled, Safety and Efficacy Trial of BHV-3000 (Rimegepant) for the Acute Treatment of Migraine
Brief Title: Safety and Efficacy in Adult Subjects With Acute Migraines
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BHV3000-302
Record Dates: First submitted 2017-07-27; First posted 2017-08-03 (Actual); Results first posted 2020-12-23 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Migraine, With or Without Aura
MeSH Terms: conditions — Migraine Disorders | interventions — rimegepant sulfate

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blind to Sponsor, Investigator and Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Rimegepant 75 mg (Experimental): Participants were administered a single oral dose of 75 mg of rimegepant tablet on occurrence of migraine that reached moderate or severe intensity up to 45 days after randomization.
  Interventions: Drug: Rimegepant
- Placebo (Placebo Comparator): Participants were administered a single oral dose of matching placebo tablet for rimegepant (75 mg) on occurrence of migraine that reached moderate or severe intensity up to 45 days after randomization.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rimegepant — 75 mg tablet QD
  Other Names: BHV-3000
  Arms: Rimegepant 75 mg
Drug: Placebo — Placebo tablet to match rimegepant dose QD
  Arms: Placebo

SUMMARY:
The purpose of this study is to compare the efficacy of BHV-3000 (rimegepant) versus placebo in subjects with Acute Migraines

ELIGIBILITY:
Key Inclusion Criteria:

1. Patient has at least 1 year history of migraines (with or without aura), consistent with a diagnosis according to the International Classification of Headache Disorder, 3rd Edition, Beta version[1] including the following:

   * Not more than 8 attacks of moderate or severe intensity per month within last 3 months
   * Consistent migraine headaches of at least 2 migraine headache attacks of moderate or severe intensity in each of the 3 months prior to the Screening Visit and maintains this requirement during the Screening Period
2. Less than 15 days with headache (migraine or non-migraine) per month in each of the 3 months prior to the Screening Visit and maintains this requirement during the Screening Period
3. Patients on prophylactic migraine medication are permitted to remain on therapy provided they have been on a stable dose for at least 3 months prior to study entry.
4. Patients with contraindications for use of triptans may be included provided they meet all other study entry criteria.

Key Exclusion Criteria:

1. Patient history of HIV disease
2. Patient history with current evidence of uncontrolled, unstable or recently diagnosed cardiovascular disease, such as ischemic heart disease, coronary artery vasospasm, and cerebral ischemia. Patients with Myocardial Infarction (MI), Acute Coronary Syndrome (ACS),Percutaneous Coronary Intervention (PCI), cardiac surgery, stroke or transient ischemic attack (TIA) during the 6 months prior to screening.
3. Uncontrolled hypertension (high blood pressure), or uncontrolled diabetes (however patients can be included who have stable hypertension and/or diabetes for 3 months prior to being enrolled)
4. Patient has a current diagnosis of major depression, other pain syndromes, psychiatric conditions (eg, schizophrenia), dementia, or significant neurological disorders (other than migraine) that, in the Investigator's opinion, might interfere with study assessments
5. Patient has a history of gastric, or small intestinal surgery, or has a disease that causes malabsorption.
6. The patient has a history or current evidence of any significant and/or unstable medical conditions (eg, history of congenital heart disease or arrhythmia, known suspected infection, hepatitisB or C, or cancer) that, in the investigator's opinion, would expose them to undue risk of a significant adverse event (AE) or interfere with assessments of safety or efficacy during the course ofthe trial
7. History of, treatment for, or evidence of, alcohol or drug abuse within the past 12 months or patients who have met DSM-V criteria for any significant substance use disorder within thepast 12 months from the date of the screening visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1499 (Actual)
Dates: Start 2017-07-27 (Actual); Primary Completion 2018-01-25 (Actual); Study Completion 2018-01-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (49):
- United States (49):
  - Coastal Clinical Research, Mobile, Alabama
  - Thunderbird Internal Medicine / Radiant Research, Inc., Glendale, Arizona
  - Woodland Research Northwest, LLC, Rogers, Arkansas
  - eStudySite, La Mesa, California
  - Collaborative Neuroscience Network, LLC, Long Beach, California
  - Pharmacology Research Institute, Los Alamitos, California
  - Pharmacology Research Institute, Newport Beach, California
  - Pacific Research Partners LLC, Oakland, California
  - National Research Institute, Panorama City, California
  - California Neuroscience Research Medical Group, Inc., Sherman Oaks, California
  - Clinical Trials of the Rockies, Denver, Colorado
  - AGA Clinical Trials, Hialeah, Florida
  - Clinical Neuroscience Solutions, Jacksonville, Florida
  - Renstar Medical Research, Ocala, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Meridien Research, Tampa, Florida
  - Radiant Research, Inc., Atlanta, Georgia
  - Savannah Neurology Specialists, Savannah, Georgia
  - Christie Clinic, LLC, Champaign, Illinois
  - PMG Research of McFrland Clinic, Ames, Iowa
  - Heartland Research Associates, LLC, Augusta, Kansas
  - Heartland Research Associates, LLC, Newton, Kansas
  - Heartland Research Associates, LLC, Park City, Kansas
  - Heartland Research Associates, LLC, Wichita, Kansas
  - MedPharmics, LLC, Metairie, Louisiana
  - NECCR Primacare Research, LLC, Fall River, Massachusetts
  - Albuquerque Neuroscience, Inc., Albuquerque, New Mexico
  - Radiant Research, Inc., Jamaica, New York
  - PMG Research of Raleigh, Inc., Raleigh, North Carolina
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - PMG Research of Wilmington, LLC, Wilmington, North Carolina
  - Radiant Research, Inc., Cincinnati, Ohio
  - Radiant Research, Inc., Columbus, Ohio
  - Midwest Clinical Research Center, Dayton, Ohio
  - Neurology Diagnostics, Inc., Dayton, Ohio
  - Aventiv Research, Inc., Dublin, Ohio
  - Summit Research Network (Oregon), Inc., Portland, Oregon
  - Oregon Center for Clinical Investigations, Inc, Salem, Oregon
  - Fieve Clinical Research, Inc., Scranton, Pennsylvania
  - Radiant Research, Inc., Anderson, South Carolina
  - Clinical Research Associates, Inc., Nashville, Tennessee
  - Tekton Research, Austin, Texas
  - Ventavia Research Group, Fort Worth, Texas
  - Red Star Research, Lake Jackson, Texas
  - FMC Science, Lampasas, Texas
  - PCP for Life, Magnolia, Texas
  - Research Across America, Mesquite, Texas
  - Doctors of Internal Medicine, LTD / Radiant Research, Inc., Plano, Texas
  - DM Clinical Research, Tomball, Texas

REFERENCES:
- [Derived] Charleston L 4th, Armand CE, Monteith TS, O'Brien HL, Abbott CC, Pixton GC, Fullerton T. Efficacy and safety of rimegepant for the acute treatment of migraine in Black or African American adults: A post hoc pooled subgroup analysis from three randomized, placebo-controlled clinical trials. Headache. 2026 Feb 6. doi: 10.1111/head.70034. Online ahead of print. PMID 41652666
- [Derived] Lipton RB, Blumenfeld A, Jensen CM, Croop R, Thiry A, L'Italien G, Morris BA, Coric V, Goadsby PJ. Efficacy of rimegepant for the acute treatment of migraine based on triptan treatment experience: Pooled results from three phase 3 randomized clinical trials. Cephalalgia. 2023 Feb;43(2):3331024221141686. doi: 10.1177/03331024221141686. PMID 36739511
- [Derived] Lipton RB, Croop R, Stock EG, Stock DA, Morris BA, Frost M, Dubowchik GM, Conway CM, Coric V, Goadsby PJ. Rimegepant, an Oral Calcitonin Gene-Related Peptide Receptor Antagonist, for Migraine. N Engl J Med. 2019 Jul 11;381(2):142-149. doi: 10.1056/NEJMoa1811090. PMID 31291516

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 50 sites in United States of which 49 sites enrolled at least 1 participant.
Pre-assignment Details: A total of 1499 participants were enrolled, of which 1186 participants were randomized to rimegepant 75 milligram (mg) or placebo. A total of 313 participants failed screening mainly due to failure to meet eligibility criteria. The randomization was stratified in a 1:1 ratio based on use of prophylactic migraine medications (yes or no).
Period: Overall Study
Arm/Group | Rimegepant 75 mg | Placebo
Started (Randomized) | 594 | 592
Treated | 543 | 543
Completed | 538 | 542
Not Completed | 56 | 50
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 13 | 10
Not completed — Not Experienced Moderate/Severe Migraine | 26 | 31
Not completed — Non-Compliance With Study Treatment | 0 | 1
Not completed — Physician Decision | 1 | 2
Not completed — Pregnancy | 1 | 0
Not completed — Protocol Deviation | 0 | 1
Not completed — Technical Problems | 8 | 1
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Other Reasons | 4 | 0

BASELINE CHARACTERISTICS:
Population: The analysis was performed on modified intent to treat (mITT) participants, defined as those who were randomized only once, took study medication, had moderate to severe pain level at migraine onset, and who provided at least 1 post-dose efficacy measurement (i.e., after taking study medication).
Groups:
- Total: Total of all reporting groups
Arm/Group | Rimegepant 75 mg | Placebo | Total
Number analyzed (Participants) | 537 | 535 | 1072
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.195 (11.8693) | 40.910 (12.1168) | 40.552 (11.9932)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 479 | 472 | 951
  Male | 58 | 63 | 121
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 77 | 83 | 160
  Not Hispanic or Latino | 460 | 452 | 912
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 5 | 9
  Asian | 8 | 8 | 16
  Native Hawaiian or Other Pacific Islander | 6 | 0 | 6
  Black or African American | 111 | 118 | 229
  White | 394 | 399 | 793
  More than one race | 14 | 5 | 19
  Unknown or Not Reported | 0 | 0 | 0
Primary Migraine Type [Count of Participants; unit: Participants]
  Migraine without Aura | 355 | 366 | 721
  Migraine with Aura | 182 | 169 | 351
Randomization Strata, Prophylactic Migraine Medication Use [Count of Participants; unit: Participants]
  Yes | 89 | 89 | 178
  No | 448 | 446 | 894

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Freedom From Pain at 2 Hours Post-dose
Description: Pain levels were assessed on a 4-point scale (none, mild, moderate, severe) using the electronic diary (eDiary). Pain freedom was defined as pain level of none.
Time Frame: 2 Hours post-dose
Population: The analysis was performed on modified intent to treat (mITT) participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Rimegepant 75 mg | Placebo
Number analyzed (Participants) | 537 | 535
Percentage of participants | 19.6 [16.2 to 22.9] | 12.0 [9.2 to 14.7]
Statistical Analysis 1: Comparison: Rimegepant 75 mg vs Placebo; Test type: Superiority; p = 0.0006, Cochran-Mantel-Haenszel; Risk Difference (RD) = 7.6, 95% CI 2-sided [3.3 to 11.9]

2. Primary Outcome: Percentage of Participants With Freedom From Most Bothersome Symptom (MBS) at 2 Hours Post-dose
Description: MBS was reported as nausea, photophobia, or phonophobia at migraine onset using the eDiary. Symptom status (absent, present) was assessed post-dose using the eDiary separately for nausea, photophobia, and phonophobia. Freedom from MBS was defined as MBS reported at onset that was absent post-dose.
Time Frame: 2 Hours
Population: The analysis was performed on mITT participants.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Rimegepant 75 mg | Placebo
Number analyzed (Participants) | 537 | 535
Percentage of Participants | 37.6 [33.5 to 41.7] | 25.2 [21.6 to 28.9]
Statistical Analysis 1: Comparison: Rimegepant 75 mg vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 12.4, 95% CI 2-sided [6.9 to 17.9]

3. Secondary Outcome: Percentage of Participants With Freedom From Photophobia at 2 Hours Post-dose
Description: Photophobia (sensitivity to light) status was measured as absent or present in the eDiary. Freedom from photophobia was defined as photophobia absent.
Time Frame: 2 hours post-dose
Population: The analysis was performed on mITT participants with photophobia present at migraine onset.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Rimegepant 75 mg | Placebo
Number analyzed (Participants) | 489 | 477
Percentage of Participants | 37.4 [33.1 to 41.7] | 22.3 [18.6 to 26.0]
Statistical Analysis 1: Comparison: Rimegepant 75 mg vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 15.1, 95% CI 2-sided [9.4 to 20.8]

4. Secondary Outcome: Percentage of Participants With Freedom From Phonophobia at 2 Hours Post-dose
Description: Phonophobia (sensitivity to sound) status was measured as absent or present in the eDiary. Freedom from phonophobia was defined as phonophobia absent.
Time Frame: 2 hours post-dose
Population: The analysis was performed on mITT participants with phonophobia present at migraine onset.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Rimegepant 75 mg | Placebo
Number analyzed (Participants) | 362 | 374
Percentage of Participants | 36.7 [31.7 to 41.7] | 26.8 [22.3 to 31.3]
Statistical Analysis 1: Comparison: Rimegepant 75 mg vs Placebo; Test type: Superiority; p = 0.0039, Cochran-Mantel-Haenszel; Risk Difference (RD) = 9.9, 95% CI 2-sided [3.2 to 16.6]

5. Secondary Outcome: Percentage of Participants With Pain Relief at 2 Hours Post-dose
Description: Pain levels were assessed on a 4-point scale (none, mild, moderate, severe) using the eDiary. Pain relief was defined as pain level of none or mild.
Time Frame: 2 hours post-dose
Population: The analysis was performed on mITT participants..
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Rimegepant 75 mg | Placebo
Number analyzed (Participants) | 537 | 535
Percentage of Participants | 58.1 [53.9 to 62.3] | 42.8 [38.6 to 47.0]
Statistical Analysis 1: Comparison: Rimegepant 75 mg vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 15.3, 95% CI 2-sided [9.4 to 21.2]

6. Secondary Outcome: Percentage of Participants With Freedom From Nausea at 2 Hours Post-dose
Description: Nausea status was measured as absent or present in the eDiary. Freedom from nausea was defined as nausea absent.
Time Frame: 2 hours post-dose
Population: The analysis was performed on mITT participants with nausea present at migraine onset.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Rimegepant 75 mg | Placebo
Number analyzed (Participants) | 355 | 336
Percentage of Participants | 48.1 [42.9 to 53.3] | 43.3 [38.0 to 48.6]
Statistical Analysis 1: Comparison: Rimegepant 75 mg vs Placebo; Test type: Superiority; p = 0.2084, Cochran-Mantel-Haenszel — P-Value ≥ 0.05; therefore, all secondary outcome measures listed after this outcome measure in the hierarchy were not tested; Risk Difference (RD) = 4.8, 95% CI 2-sided [-2.7 to 12.2]

7. Secondary Outcome: Percentage of Participants With Rescue Medication Use Within 24 Hours Post-dose
Description: Participants who did not experience relief of their migraine headache at the end of 2 hours after dosing with study medication (and after the 2-hour assessments had been completed on the eDiary) were permitted to use the following rescue medications: aspirin, ibuprofen, acetaminophen up to 1000 mg/day (this includes Excedrin Migraine), naproxen (or any other type of nonsteroidal anti-inflammatory drug), antiemetics (e.g., metoclopramide or promethazine), or baclofen. The participant's use of rescue medication was recorded by the participant in a paper diary.
Time Frame: 24 hours post-dose
Population: The analysis was performed on mITT participants.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Rimegepant 75 mg | Placebo
Number analyzed (Participants) | 537 | 535
Percentage of Participants | 21.0 [17.6 to 24.5] | 37.0 [32.9 to 41.1]

8. Secondary Outcome: Percentage of Participants With Sustained Pain Freedom From 2 to 24 Hours Post-dose
Description: Pain levels were assessed on a 4-point scale (none, mild, moderate, severe) using the eDiary. Sustained pain freedom was defined as pain level of none at 2 hours up to 24 hours post-dose with no rescue medication use through 24 hours post-dose.
Time Frame: From 2 hours up to 24 hours post-dose
Population: The analysis was performed on mITT participants
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Rimegepant 75 mg | Placebo
Number analyzed (Participants) | 537 | 535
Percentage of Participants | 12.3 [9.5 to 15.1] | 7.1 [4.9 to 9.3]

9. Secondary Outcome: Percentage of Participants With Sustained Pain Relief From 2 to 24 Hours Post-dose
Description: Pain levels were assessed on a 4-point scale (none, mild, moderate, severe) using the eDiary. Sustained pain relief was defined as pain level of none or mild at 2 hours up to 24 hours post-dose with no rescue medication use through 24 hours post-dose.
Time Frame: From 2 hours up to 24 hours post-dose
Population: The analysis was performed on mITT participants.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Rimegepant 75 mg | Placebo
Number analyzed (Participants) | 537 | 535
Percentage of Participants | 42.6 [38.5 to 46.8] | 26.5 [22.8 to 30.3]

10. Secondary Outcome: Percentage of Participants With Sustained Pain Freedom From 2 to 48 Hours Post-dose
Description: Pain levels were assessed on a 4-point scale (none, mild, moderate, severe) using the eDiary. Sustained pain freedom was defined as pain level of none at 2 hours up to 48 hours post-dose with no rescue medication use through 48 hours post-dose.
Time Frame: From 2 hours up to 48 hours post-dose
Population: The analysis was performed on mITT participants.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Rimegepant 75 mg | Placebo
Number analyzed (Participants) | 537 | 535
Percentage of Participants | 9.9 [7.3 to 12.4] | 6.0 [4.0 to 8.0]

11. Secondary Outcome: Percentage of Participants With Sustained Pain Relief From 2 to 48 Hours Post-dose
Description: Pain levels were assessed on a 4-point scale (none, mild, moderate, severe) using the eDiary. Sustained pain relief was defined as pain level of none or mild at 2 hours up to 48 hours post-dose with no rescue medication use through 48 hours post-dose.
Time Frame: From 2 hours up to 48 hours post-dose
Population: The analysis was performed on mITT participants.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Rimegepant 75 mg | Placebo
Number analyzed (Participants) | 537 | 535
Percentage of Participants | 36.3 [32.2 to 40.4] | 22.6 [19.1 to 26.2]

12. Secondary Outcome: Percentage of Participants With Pain Relapse From 2 to 48 Hours Post-dose
Description: Pain levels were assessed on a 4-point scale (none, mild, moderate, severe) using the eDiary. Pain relapse was defined as pain level of mild, moderate, or severe after 2 hours up to 48 hours for the participants who were pain-free at 2 hours post-dose.
Time Frame: From 2 hours up to 48 hours post-dose
Population: The analysis population was performed on mITT participants with pain freedom at 2 hours post-dose.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Rimegepant 75 mg | Placebo
Number analyzed (Participants) | 105 | 64
Percentage of Participants | 49.6 [40.1 to 59.1] | 50.0 [37.8 to 62.1]

13. Secondary Outcome: Percentage of Participants With Freedom From Functional Disability at 2 Hours Post-dose
Description: Functional disability level was assessed in the eDiary on a 4-point scale: normal function, mild impairment, severe impairment, required bed rest. Freedom from functional disability was defined as normal function.
Time Frame: 2 hours post-dose
Population: The analysis was performed on mITT participants.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Rimegepant 75 mg | Placebo
Number analyzed (Participants) | 537 | 535
Percentage of Participants | 32.6 [28.6 to 36.5] | 23.4 [19.8 to 26.9]

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) were collected from informed consent up to the end of the study, and adverse events (AEs) were collected from randomization up to end of the study (up to 52 days).
Description: The safety population, all enrolled participants who received at least 1 dose of rimegepant or placebo, was used to determine the number of participants at risk for SAEs and other AEs.
Arm/Group | Rimegepant 75 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/543 | 0/543
Serious Adverse Events (participants affected / at risk) | 1/543 | 2/543
Other Adverse Events (participants affected / at risk) | 0/543 | 0/543
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rimegepant 75 mg (N=543) | Placebo (N=543)
Chest Pain (General disorders) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-01-23): https://cdn.clinicaltrials.gov/large-docs/45/NCT03237845/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-20): https://cdn.clinicaltrials.gov/large-docs/45/NCT03237845/SAP_001.pdf